CLINICAL TRIAL: NCT01778816
Title: Calf Muscle Atrophy After Achilles Tendon Rupture. A Clinical-Radiological-Biomechanical Multicenter Study.
Status: Completed | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Collaborators: Hospital Fribourg, Switzerland (Unknown); Hospital Liestal, Switzerland (Unknown)
Responsible Party: Principal Investigator, Claudio Rosso, Claudio Rosso MD MSc, University Hospital, Basel, Switzerland
Other Study IDs: RossoAchilles
Record Dates: First submitted 2013-01-25; First posted 2013-01-29 (Estimated); Last update posted 2013-01-29 (Estimated); Status verified 2013-01

CONDITIONS: Achilles Tendon Ruptures
Keywords: Achilles tendon, muscle volume, Achilles tendon length, force, ATRS, Hannover, AOFAS

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Multicenter Achilles tendon study Switzerland. Comparing three mainstream treatment types: open, percutaneous and conservative (non-operative) treatments.

Comparing force torque measurements, muscle volume and clinical scores.

ELIGIBILITY:
Inclusion Criteria:

* 20-65 years of age,
* a healthy, contralateral leg
* physiological, clinically determined alignment of the knee, foot and ankle
* no trauma to the healthy leg
* no neuromuscular impairments including muscle dystrophies
* no other posttraumatic injuries or osteoarthritis of the knee, foot or ankle of the affected leg.

Exclusion Criteria:

* re-rupture or reoperation of the Achilles tendon
* surgical site infection
* neuromuscular diseases including muscle dystrophies
* ankle valgus of more than 15° or ankle varus of more than 5°
* other known pathologies of the non-affected leg
* general MRI exclusion criteria (e.g. pacemaker, other metal not qualifying for an MRI, tattoos and claustrophobia)
* body mass index (BMI) of > 40 kg/m2

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: * Age 20-65 years
  * BMI < 40
  * no injury to leg
  * no injury on contralateral leg
Sampling Method: Probability Sample
Enrollment: 52 (Actual)
Dates: Start 2009-01; Primary Completion 2009-07 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Muscle Volume | at least 3 years after injury